CLINICAL TRIAL: NCT05293717
Title: Topical Ruxolitinib (Jak1/Jak2 Inhibitor) in Chronic Hand Dermatitis Attenuates Inflammation and Enhances Skin Barrier Repair
Brief Title: Topical Ruxolitinib in Chronic Hand Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Anna De Benedetto, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006638
Record Dates: First submitted 2022-03-07; First posted 2022-03-24 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hand Dermatitis
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All Participants (Experimental): You are being asked to apply topical medication called Ruxolitinib cream to your skin at home twice daily.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — 1.5% Ruxolitinib cream

SUMMARY:
This is an investigator-initiated, proof of concept, open study to assess efficacy of a topical Ruxolitinib in subjects with Chronic Hand Dermatitis (CHD). The study will be conducted at the University of Rochester Medical center, Dermatology Department - Rochester, NY. Qualified and enrolled subjects (see Inclusion/Exclusion criteria) will be required to come to URMC Dermatology Clinic for at least five visits.

DETAILED DESCRIPTION:
This is a single-center study anticipating to enroll 15 participants with chronic hand dermatitis. Eligible participants will receive Ruxolitinib to apply twice daily for 12 weeks. Participants will be required to be seen every 4 weeks until week 16.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hand eczema defined as hand eczema, which has persisted for more than 3 months or returned twice or more within the last 12 months.
* Disease severity graded as moderate to severe according to IGA (i.e., IGA ≥2).
* Recent history (within 1 year before the screening visit) of inadequate response to topical corticosteroid and/or calcineurin inhibitors treatment or topical corticosteroid treatment being medically inadvisable.

Exclusion Criteria:

* Active atopic dermatitis in regions other than the hands requiring medical treatment.
* Active psoriasis in regions other than the hands requiring medical treatment.
* Clinically significant infection (e.g., impetiginized hand eczema or tinea manum) on the hands.
* Patients with excessive contact of hands with water (longer than 2 hours at day; or > 20 hands washing at day) that is believed to be a predominant cause of the hand dermatitis.
* Subjects with known antigen sensitization based on Patch test (with 3 years) that are unable to reduce contact with the specific antigen(s).
* Subjects chronically and consistently exposed to known-irritant or other substance known to impact skin barrier will be excluded based on PI judgement
* Systemic treatment with immunosuppressive drugs, immunomodulating drugs, retinoids, or corticosteroids within 4 weeks prior to baseline.
* Systemic treatment with antibiotics within 4 weeks prior to baseline
* Phototherapy on the hands within 4 weeks prior to baseline.
* Use of topical immunomodulators (e.g., phosphodiesterase-4 (PDE-4) inhibitors, pimecrolimus, tacrolimus) or topical corticosteroids on the hands within 2 weeks prior to baseline.
* Use of topical antibiotics on the hands within 2 weeks prior to baseline.
* Change in systemic antihistamine therapy within 2 weeks prior to baseline i.e., subjects must not start antihistamine treatment or change the current dosage regime within 2 weeks prior to baseline.
* Other topicals applied therapy on the hands (except for the use of subject's own emollients) within 1 week prior to baseline.
* Receipt of any marketed or investigational biologic agents within 6 months or 5 half-lives prior to baseline
* Any disorder which is not stable and in the investigator's opinion could affect the safety of the subject, influence the findings of the trial, or impede the subject's ability to complete the trial.
* Participants with clinically significant cytopenia at screening
* Participants with severely impaired liver or kidney function and unstable.
* Participants who have previously received JAK inhibitor therapy, systemic or topical.
* History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV), or the subject taking antiretroviral medications.
* Females who are breastfeeding, pregnant, or anticipate becoming pregnant during the study time frame
* History of skin cancer on hands within 5 years.
* History of recalcitrant warts on hands within 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UR Medicine Dermatology College Town, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 subjects were consented but 4 failed screening leaving 16 participants who started the intervention
Period: Overall Study
Arm/Group | All Participants
Started | 16
Completed | 15
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Duration of chronic hand dermatitis (CHD) [Mean (Standard Deviation); unit: years] | 7.5 (8.8)
mean Hand Eczema Severity Index [Mean (Standard Deviation); unit: units on a scale] — Hand Eczema Severity Index (HECSI) , a well-accepted and validated scoring system for disease activity. It incorporates both the extent and the intensity of the disease. Each hand is divided into five areas: fingertips, fingers (except the tips), palms, back of hands and wrists. Each area will be scored for extension and intensity of the six following clinical signs: erythema, induration ⁄papulation, vesicles, fissuring, scaling and edema; which are graded on the following scale: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe. The score ranges from 0-360.
  units on a scale | 56.2 (24.2)
Number of participants with atopic CHD subtype [Number; unit: participants] | 7
number of participants with hyperkeratotic morphology [Number; unit: participants] | 7
number of participants with recurrent vesicular morphology [Number; unit: participants] | 1
number of participants with mixed morphology [Count of Participants; unit: Participants] | 1
number of participants who previously attempted taking CHD therapy [Count of Participants; unit: Participants]
  high-potency topical steroids | 16
  tacrolimus | 4
  methotrexate | 3
  oral steroids | 3
  mycophenolate | 1
  phototherapy | 3
  calcipotriene | 1
  acitretin | 3
number of participants with an Investigators Global Assessment (IGA) score of 3 or more [Count of Participants; unit: Participants] — The Investigator Global Assessment (IGA) will provide information of the overall disease. It is a 5-point scale: 1-clear, 2-almost clear, 3-mild, 4-moderate and 5-severe.
  Participants
    IGA-3 | 8
    IGA-4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Chronic Hand Dermatitis Improvement as Assessed by Investigators Global Assessment
Description: Proportion of patients achieving an Investigators Global Assessment (IGA) score of 0 or 1 with at least a 2-step improvement (IGA treatment success). The Investigator Global Assessment (IGA) will provide information of the overall disease. It is a 5-point scale: clear-1, almost clear-2, mild-3, moderate-4, and severe-5.
Time Frame: week 12
Measure: Number; unit: proportion of participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
proportion of participants | 0.53

2. Primary Outcome: Percent Change in Mean Hand Eczema Severity Index (HECSI)
Description: Hand Eczema Severity Index (HECSI) , a well-accepted and validated scoring system for disease activity. It incorporates both the extent and the intensity of the disease. Each hand is divided into five areas: fingertips, fingers (except the tips), palms, back of hands and wrists. Each area will be scored for extension and intensity of the six following clinical signs: erythema, induration /papulation, vesicles, fissuring, scaling, and edema; which are graded on the following scale: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe. Data will be reported as a percent change in the HECSI score from baseline to week 12. The score ranges from 0-360.
Time Frame: baseline to week 12
Measure: Mean (Standard Error); unit: percent change of HECSI index
Arm/Group | All Participants
Number analyzed (Participants) | 15
percent change of HECSI index | -86.2 (3.72)
Statistical Analysis 1: Comparison: All Participants; Test type: Other — This is an open-label study. No power calculation was performed; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=16)
kidney stone (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=16)
Upper Respiratory Infection (Infections and infestations) | 1
scalp abscess (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT05293717/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT05293717/ICF_001.pdf